CLINICAL TRIAL: NCT01655745
Title: LCCC 1209: Pilot Study of [18F] Fluorodeoxyglucose Positron Emission Tomography-Magnetic Resonance Imaging (FDG-PET-MRI) for Staging of Muscle-Invasive Bladder Cancer
Brief Title: Positron Emission Tomography (PET) Study for Staging of Muscle Invasive Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1209
Record Dates: First submitted 2012-07-26; First posted 2012-08-02 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Bladder Cancer
Keywords: [18F]; FDG Positron Emission Tomography-Magnetic Resonance Imaging; FDG-PET-MRI; Muscle-Invasive Bladder Cancer; Pilot Study; LCCC 1209; UNC Lineberger; MDCT
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FDG PET/MR, No Chemotherapy Arm (Experimental): Patients that are NOT receiving chemotherapy but are only completing surgical intervention.
  Interventions: Procedure: FDG PET/MR
- FDG PET/MR, Chemotherapy Arm (Experimental): Patients that are receiving chemotherapy prior to completing surgical intervention. These patients will receive a FDG PET/MR prior to chemotherapy and after completion of chemotherapy (at the time of pre-op, before surgical intervention).
  Interventions: Procedure: FDG PET/MR

INTERVENTIONS:
Procedure: FDG PET/MR — All patients will undergo a gadolinium enhanced MRI with simultaneous acquisition of FDG-PET prior to planned radical cystectomy and pelvic lymph node dissection
  Other Names: Fluorodeoxyglucose Positron Emission Tomography MRI

SUMMARY:
This prospective pilot study will enroll 30 patients with cT2/T3-N0-M0 urothelial carcinoma of the bladder for whom radical cystectomy with pelvic lymph node dissection is planned. This pilot study is designed to provide preliminary information on the accuracy of [18F] Fluorodeoxyglucose Positron Emission Tomography MRI (FDG-PET-MRI) in the staging of muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
This prospective pilot study will enroll 30 patients with cT2/T3-N0-M0 urothelial carcinoma of the bladder for whom radical cystectomy with pelvic lymph node dissection is planned. This pilot study is designed to provide preliminary information on the accuracy of [18F] Fluorodeoxyglucose Positron Emission Tomography MRI (FDG-PET-MRI) in the staging of muscle-invasive bladder cancer. All patients will undergo baseline FDG-PET-MRI and routine (standard of care) contrast enhanced abdominal/pelvic multi-detector computed tomography (MDCT). The imaging results will ultimately be compared to final pathology as the gold standard. If the accuracy of FDG-PET-MRI is improved as compared to standard MDCT, the investigators plan to conduct a larger follow-up study to confirm the results of this pilot study. In addition, this pilot study will set the stage for the evaluation of novel PET tracers in the imaging of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age (no upper age limit)
* Informed consent obtained and signed
* cT2/T3-N0-M0 urothelial carcinoma of the bladder
* Planned radical cystectomy with pelvic lymph node dissection
* No known local regional or distant metastatic disease
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to FDG-PET-MRI

Exclusion Criteria:

* History of severe reaction to contrast-enhanced CT scan
* Poorly controlled diabetes mellitus
* Inability to tolerate PET and/or MRI
* Presence of pacemaker or intracranial aneurysm clip
* Serum creatinine >1.8 mg/dL OR GFR < 30mL/min
* Pregnant or lactating female
* Inability to lie flat for >1 hour
* Body Mass Index (BMI) >35
* History of a prior malignancy within past 5 years are excluded unless they have been disease free for 3 or more years or unless they have a completely resected non-melanoma skin cancer.
* Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the FDG-PET-MRI for staging of muscle-invasive bladder cancer | 3 years
  The sensitivity and specificity of the FDG-PET-MRI for staging of muscle-invasive bladder will be evaluated by using the pathology from the radical cystectomy and lymph node dissection specimen or biopsy as the reference standard. The sensitivity and specificity of FDG-PET-MRI will be compared to conventional CT performed in all patients in this pilot study and FDG-PET-CT.

SECONDARY OUTCOMES:
Association of FDG-PET-MRI with RFS, DSS and OS in patients with muscle-invasive bladder cancer | 3 years
  A positive FDG-PET-MRI or routine contrast enhanced abdominal/pelvic MDCT will be defined as evidence of metastatic disease as follows: 1) regionally, in the pelvic lymph nodes; or 2) distantly, to bone, lung, viscera or lymph nodes outside of the pelvis. OS will be defined as the time from the PET-MRI to the date of death from any cause. DSS will be defined from the date of PET-MRI to the date of death from disease. RFS will be defined as the time from the date of PET-MRI to recurrence or death from disease.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew I. Milowsky, MD, Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: National Cancer Institute (NCI) website — http://www.cancer.gov/